CLINICAL TRIAL: NCT04595851
Title: Implementation of a Model Integrating Primary and Oncology Care for Patients Taking Oral Anticancer Agents (OAA)
Brief Title: Pharmacists Coordinated Care Oncology Model (PCOM) for Patients Taking Oral Anti-cancer Medications
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: accrual difficulties
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UMCC 2020.053; HUM00178781 (Other: University of Michigan)
Record Dates: First submitted 2020-10-13; First posted 2020-10-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Chronic Myeloid Leukemia; Chronic Lymphocytic Leukemia; Multiple Chronic Conditions
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Chronic Conditions | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacist Coordinated care Oncology Model (PCOM) (Other): The Pharmacist Coordinated care Oncology Model includes patient self-reported symptoms and medication adherence, comprehensive medication review(s) and intentional communication between oncology and primary care pharmacists.
  Interventions: Other: Patient Reported Outcome Measure (PROM); Other: Comprehensive Medication Review (CMR); Other: Communications between oncology and primary care pharmacists

INTERVENTIONS:
Other: Patient Reported Outcome Measure (PROM) — Participants will complete a PROM (Michigan Oncology Quality Consortium, Patient Assessment Tool for Oral Chemotherapy) for their oral anticancer agent (OAA) at two timepoints over 2 months, to assess patient symptoms and adherence to OAA.
Other: Comprehensive Medication Review (CMR) — Following the first PROM, participants will be contacted by the primary care pharmacist for a Comprehensive Medication Review (CMR) for their chronic medications. If warranted, a follow-up CMR will take place after the second PROM.
Other: Communications between oncology and primary care pharmacists — Throughout the study, the oncology and primary care pharmacists will communicate about medications through the electronic medical record.

SUMMARY:
The objective of this study is to improve medication, symptom, and disease management of patients with hematological malignancies and multiple chronic conditions (2 or more conditions in addition to cancer) through care coordination between pharmacists working in oncology practices and those working in primary care practices (Pharmacists Coordinated care Oncology Model [PCOM]).

This is a pilot study in which the investigators will examine the association between outcome measures, but the study design and sample size are insufficient to quantify the impact of OAA initiation or OAA adherence on adherence to chronic medications. This pilot study and data analyses are being done in preparation for a larger, controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Has primary care physician
* Diagnosis of chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), chronic myeloid leukemia (CML), or multiple myeloma (MM)
* Initiating an OAA, either for the first time or a change from previous OAA
* Diagnosis of at least 2 chronic conditions, including at least one of the following: diabetes, hypertension, hyperlipidemia, congestive heart failure, depression/anxiety, gastroesophageal reflux disease, and/or chronic obstructive pulmonary disease
* Patients taking at least two chronic medications, including at least one medication for one of the conditions listed above.
* Willing and able to sign informed consent.

Exclusion Criteria:

* Cannot speak English
* Concurrent diagnosis of type 1 diabetes
* Concurrent diagnosis of human immunodeficiency virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Dose-adjusted proportion of days covered (PDC) for oral anti-cancer agent (OAA) | Up to 6 months following OAA initiation
  PDC is a common way to assess a patient's adherence to a medication regimen. PDC is the ratio of number of days the patient is supplied with OAA medication, from the time of OAA initiation until 6 months later, to the total number of days during that period. For OAAs, data from the electronic medical record (EMR) for dose changes will be aligned with the refill data to calculate a dose-adjusted PDC.
PDC for chronic condition medications | Up to 6 months following OAA initiation
  PDC is the ratio of the number of days the patient is supplied with chronic condition medications, from the time of OAA initiation until 6 months later, to the total number of days during that period.

SECONDARY OUTCOMES:
Percent of patients with two completed Patient Reported Outcome Measures (PROMs) | Up to day 42 (+/-3) after OAA initiation
  The Michigan Oncology Quality Consortium (MOQC) OAA PROM, Patient Assessment Tool for Oral Chemotherapy is to be completed at 2 and 6 weeks after OAA initiation. This measure assesses the percent of patients who complete this PROM at both time points.
Percent of patients with completed Comprehensive Medication Reviews (CMRs) | Day 50 (+/-3) after OAA initiation
  Completed CMR includes initial and follow-up CMR with primary care pharmacist.
Percent of patients with scheduled Comprehensive Medication Review (CMR) within one week of first PROM result | Day 22 (+/-3) after OAA initiation
  The PROM is scored within one day after it is completed by the patient. The primary care pharmacist sets a date and time for the initial CMR after receiving the first scored PROM.
Percent of patients where oncology pharmacist reviewed PROM within 1 day of receiving scored PROM | Up to day 44 (+/-3) after OAA initiation
  The PROM is scored within one day after it is completed by the patient and is routed to the oncology pharmacist to review the results. The number of PROMs that are reviewed within 1 day of receipt will be assessed at 2 weeks and at 6 weeks.
Percent of CMRs where note was routed to oncology pharmacist | Up to day 43 (+/-3) after OAA initiation
  The number of CMR where note was routed to oncology pharmacist out of total number of completed CMRs, assessed at 2 weeks and at 6 weeks.
Percent of CMR notes that oncology pharmacist reviewed | Up to day 44 (+/-3) after OAA initiation
  The number of CMR notes reviewed by the oncology pharmacist out of the total number of completed CMRs, assessed at 2 weeks and at 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Farris, PhD, Principal Investigator — University of Michigan College of Pharmacy
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No